CLINICAL TRIAL: NCT07049874
Title: The Effect of Huel on Markers of Inflammation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: Aelius Biotech (Unknown)
Responsible Party: Principal Investigator, Anthony Watson, Lecturer in Human Nutrition, Newcastle University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Prot1
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: 4 Weeks Supplementation of Huel Ready to Eat Foods
Keywords: protein; plant based; Plant protein; inflammation
MeSH Terms: conditions — Inflammation | interventions — SLC30A9 protein, human

STUDY DESIGN:
Masking Description: This is an open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4 weeks consumption of Huel ready to eat foods (Experimental)
  Interventions: Dietary Supplement: Huel

INTERVENTIONS:
Dietary Supplement: Huel — Ready to eat huel foods. Containing 2 ready to drink shakes, one savoury meal pack and meal replacement powder. Consumption amounts were based on energy needs of each person

SUMMARY:
This project will assess the effect of Huel on markers of gastrointestinal inflammation of 30 generally healthy individuals. The aim is to identify any changes in the markers of inflammation status of volunteers in any of the 9 markers to be monitored. Inflammation status will be measured at the start of the study, after one week of their habitual diets and again after four weeks of consuming two ready to drink Huel products per day, one Hot & Savoury Huel (grain-based option only) and the remainder of their calorie intake to be made up of Huel Powder (v3.1).

ELIGIBILITY:
Inclusion Criteria:

Generally healthy Aged 18 years and over Non-pregnant, Non-lactating non-smoking

Exclusion Criteria:

Smoker Pregnant Lactating BMI >30 Food allergy Disordered eating Disorder which could impact the study outcomes Medications which could impact the study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
C-Reactive protein | baseline and after 4 weeks supplementation
neutrophils | baseline and after 4 weeks supplementation
TNF-alpha | baseline and after 4 weeks supplementation
IL-10 | baseline and after 4 weeks supplementation
IL-6 | baseline and after 4 weeks supplementation

SECONDARY OUTCOMES:
linoleic acid | baseline and after 4 weeks supplementation
arachidonic acid | baseline and after 4 weeks supplementation
alpha-linoleic acid | baseline and after 4 weeks supplementation
eicosapentaenoic acid | baseline and after 4 weeks supplementation
Body Mass Index | baseline and after 4 weeks supplementation
Body mass | baseline and after 4 weeks supplementation
Waist cercumference | baseline and after 4 weeks supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Anthony W Watson, PhD, Principal Investigator — Newcastle University
Locations (1):
- Faculty of Medical Sciences, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is not acceptable due to the ethical approval given